CLINICAL TRIAL: NCT03895112
Title: Phase I Study of AVID200 in Patients With Myelofibrosis (Myeloproliferative Neoplasms Research Consortium [MPN-RC] 118)
Brief Title: MPN-RC 118 AVID200 in Myelofibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: John Mascarenhas (Other)
Collaborators: Formation Biologics (Industry); National Cancer Institute (NCI) (NIH); Myeloproliferative Neoplasm Research Consortium (MPN-RC) (Unknown)
Responsible Party: Sponsor-Investigator, John Mascarenhas, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 07-0548-01401; P01CA108671 (NIH); MPN-RC 118 (Other: Myeloproliferative Neoplasm Research Consortium)
Record Dates: First submitted 2019-03-22; First posted 2019-03-29 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Primary Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post ET MF; Post PV MF
Keywords: Therapeutic; Fibrosis; Splenomegaly; Myeloproliferative neoplasms research consortium; Intravenous Infusion; Phase 1
MeSH Terms: conditions — Primary Myelofibrosis; Fibrosis; Splenomegaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AVID200 (Experimental): intravenous in dose cohorts of 70mg/m2 or 180 mg/m2
  Interventions: Drug: AVID200

INTERVENTIONS:
Drug: AVID200 — dose cohorts of 21-day cycles

SUMMARY:
Increased levels of TGF-β1 were detected in serum, plasma and BM and positively correlated with both grade of BMF and extent of leukemic cell infiltration in the marrow. TGF-β likely plays a dual role in promoting myelofibrosis and myeloproliferation, both of which are the bone marrow morphologic hallmark of MF. AVID200 is a drug that targets TGF-β1 and TGF-β3. The study team hypothesizes that inhibiting the TGF-β signaling pathway in MF will decrease the fibrogenic stimuli leading to myelofibrosis and concomitantly interrupt myeloproliferation and restore normal hematopoiesis.

This is a first in human, open-label, multicenter, Phase I/Ib trial of AVID200. Patients must have intermediate-2 or higher primary myelofibrosis (PMF), post-essential thrombocythemia or polycythemia-vera related MF (Post ET/PV MF). This study will enroll up to 24 patients. AVID200 is delivered by IV infusion on day 1 of each 3 week cycle.

DETAILED DESCRIPTION:
This is a first in human, open-label, multicenter, Phase I/Ib trial of AVID200. To date, there is no therapy for MF evaluated in the clinic that clearly demonstrates the ability to target the malignant HSC and result in effective and reproducible bone marrow morphologic, cytogenetic and molecular responses. Medicinal therapies that result in disease course modification are urgently needed in this chronic and progressive myeloid malignancy. TGF-β likely plays a dual role in promoting myelofibrosis and myeloproliferation, both of which are the bone marrow morphologic hallmark of MF. The study team proposes that inhibiting the TGF-β signaling pathway in MF will decrease the fibrogenic stimuli leading to myelofibrosis and concomitantly interrupt myeloproliferation and restore normal hematopoiesis. AVID200 is a fusion protein containing TGF-β receptor ectodomains fused to a human Fc IgG domain. AVID200 is a potent TGFβ trap with antibody-like properties which has pM potency against two of the three TGFβ ligands, TGFβ1 and β3.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥18 years of age at the time of signing the Informed Consent Form (ICF)
* Subjects must voluntarily sign an ICF
* Subjects must have a pathologically confirmed diagnosis of PMF as per the WHO diagnostic criteria or post ET/PV MF (note that all diagnoses must include the presence of at least Grade 2 marrow fibrosis according to the European Consensus on Grading of Bone Marrow Fibrosis (see Table 6) with intermediate -2 or high risk disease according to the IWG-MRT Dynamic International Prognostic Scoring System (DIPSS) (see Table 7)
* A bone marrow biopsy must be performed within the 30 day screening period, however, a bone marrow biopsy obtained within 90 days of screening without intervening treatments and approved by the study chair may suffice.
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
* Life expectancy of at least six months
* At least two weeks must have elapsed between the last dose of any MF-directed drug treatments (including investigational therapies and excluding hydroxyurea) and study enrollment
* Not eligible for ruxolitinib therapy due to a platelet count <50 x 109/L, previously treated and lack/loss of response as defined by at least one of the following:

  1. Treatment for ≥3 months with inadequate efficacy response defined as <10% spleen volume reduction by MRI or <30% decrease from baseline in spleen length by physical examination or regrowth to these parameters following an initial response; and/or
  2. Treatment for ≥28 days complicated by either

  i. Development of a red blood cell transfusion requirement (at least 2 units/month for 2 months) ii. National Cancer Institute (NCI) CTCAE grade ≥ 3 AEs of thrombocytopenia, anemia, hematoma, and/or hemorrhage while being treated with a dosage of < 20 mg BID
* Recovery to ≤ Grade 1 or baseline of any toxicities due to prior systemic treatments, excluding alopecia
* Women of child bearing potential (WCBP), defined as a sexually mature woman not surgically sterilized or not post-menopausal for at least 24 consecutive months if ≤55 years or 12 months if >55 years, must have a negative serum pregnancy test at screening and cycle 1 day 1 and must agree to use adequate methods of birth control throughout the study. Adequate methods of contraception include use of oral contraceptives or Depo-Provera, with an additional barrier method (diaphragm with spermicidal gel or condoms with spermicide), double-barrier methods (diaphragm with spermicidal gel and condoms with spermicide), partner vasectomy, and total abstinence.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Must have adequate organ function as demonstrated by the following:

  1. ALT (SGPT) and/or AST (SGOT) ≤ 3x upper limit of normal (ULN), or ≤ 4 x ULN (if upon judgment of the treating physician, it is believed to be due to extramedullary hematopoiesis [EMH] related to MF);
  2. Direct bilirubin ≤ 1.5 x ULN; or ≤ 2x ULN (if upon judgment of the treating physician, it is believed to be due to extra-medullary hematopoiesis related to MF or documented Gilbert's syndrome);
  3. Serum creatinine ≤ 2.0 mg/dL;
  4. Platelet count ≥25 x 109/L
* Ability to adhere to the study visit schedule and all protocol requirements
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Other invasive malignancies within the last 3 years, except non-melanoma skin cancer and localized cured prostate and cervical cancer.
* Previous exposure to galunisertib, fresolimumab, sotatercept, or luspatercept.
* History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months
* Have moderate or severe cardiovascular disease:

  1. have the presence of cardiac disease, including a myocardial infarction within 6 months prior to study entry, unstable angina pectoris, New York Heart Association Class III/IV congestive heart failure, or uncontrolled hypertension
  2. have documented major ECG abnormalities (not responding to medical treatments)
* Have predisposing conditions that are consistent with development of aneurysms of the ascending aorta or aortic stress (for example, family history of aneurysms, Marfan-Syndrome, bicuspid aortic valve, evidence of damage to the large vessels of the heart documented by CT scan/MRI with contrast)
* Presence of active serious infection;
* Any serious, unstable medical or psychiatric condition that would prevent, (as judged by the Investigator) the subject from signing the informed consent form or any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Known history of human immunodeficiency virus (HIV), or known active hepatitis A, B, or C infection
* Organ transplant recipients other than bone marrow transplant
* Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Maximally tolerated dose (MTD) of AVID200 | After 6 cycles (Each cycle is 21 days)
  Cohorts of 3 patients with a maximum evaluable sample size of 12 patients and a target toxicity rate of 30% to estimate the MTD. Each cycle is 21 days.
Number of patients with response eligibility for Phase 1b | After 6 cycles
  Subjects attaining at least a CI (clinical improvement) by IWG/ELN criteria, or a decrease in bone marrow fibrosis by ≥1 grade with otherwise stable disease, will be allowed to continue AVID200 in the extension phase of the trial.

SECONDARY OUTCOMES:
IWG/ELN criteria | After 6 cycles and after 12 cycles (Each cycle is 21 days)
  response by IWG/ELN criteria at the end of Cycle 6 and Cycle 12. The IWG/ELN criteria: CR (complete remission), PR (partial remission), Clinical improvement, Anemia response, Spleen response, Symptoms response, PD (progressive disease), SD (stable disease), Relapse, Cytogenetic remission, and Molecular remission
Bone marrow fibrosis grade | up to 37 days after 13 cycles (Each cycle is 21 days)
  bone marrow fibrosis grade at the end of Cycle 6 and 12. Bone marrow fibrosis (MF) is graded as MF-0 to MF-3, with higher number indicating more disease.
Myelofibrosis Symptom Assessment Form (MFSAF) | up to 37 days after 13 cycles (Each cycle is 21 days)
  MF-SAFv4.0,each of the items are scored 0 to 10, with total summation from 0 to 100, with higher score indicating more symptoms.
EORTC QLQ-C30 | up to 37 days after 13 cycles (Each cycle is 21 days)
  EORTC QLQ-C30, 28 item scored from 1 (not at all) to 4 (very much), and 2 items scored 1 (very poor) to 7 (excellent). Total score from 28 - 126, with higher score indicating poorer health

CONTACTS AND LOCATIONS:
Overall Officials: John Mascarenhas, MD, Study Chair — Icahn School of Medicine at Mount Sinai; Ruben Mesa, MD, Study Chair — Mays Cancer Center at UT Health; Ronald Hoffman, MD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Varricchio L, Mosoyan G, Elghaity-Beckley S, Mia MB, Handa S, Salib C, Mascarenhas J, Hoffman R. Thrombocytopenia in myelofibrosis is characterized by inflammatory megakaryocytes with reduced G6B expression. Blood. 2025 Sep 25;146(13):1612-1624. doi: 10.1182/blood.2024027363. PMID 40643151